CLINICAL TRIAL: NCT03079284
Title: The Effects of Holding on Stress and Bonding in Mother-Infant Dyads During Therapeutic Hypothermia
Brief Title: Holding, Stress, and Bonding During Therapeutic Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexa Craig (Other)
Collaborators: MaineHealth (Other)
Responsible Party: Sponsor-Investigator, Alexa Craig, Assistant Professor of Pediatrics, MaineHealth
Organization: MaineHealth (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1015281-1
Record Dates: First submitted 2017-03-06; First posted 2017-03-14 (Actual); Results first posted 2022-01-26 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Holding Group (Experimental): After meeting inclusion criteria and consenting to participation, mothers of infants who have completed at least 24 hours of therapeutic hypothermia treatment will be allowed to hold their infant who will remain on the cooling blanket for a 30-minute period with the use of a thermal barrier. Vital signs will be measured before holding begins, during holding and following completion of holding. Temperature will be recorded every two minutes during holding. Afterwards, a Likert scale questionnaire to assess the mother's and nurse's reactions will be administered.
  Interventions: Other: Holding during cooling

INTERVENTIONS:
Other: Holding during cooling — An initial set of vital sings will be recorded before the infant is removed from the isolette. The mother will sit in a reclining chair next to the isolette and place a thermal barrier over her chest and abdomen. The infant will be transferred to the mother by placing the hands under the cooling blanket so as to move the infant and cooling blanket together as one unit. The mother will be allowed to hold for thirty minutes provided that the infant's temperature does not increase by greater than one degree centigrade and the oxygen saturation does not drop below 90%. After thirty minutes, the infant will be returned to the isolette.

SUMMARY:
Ten infants undergoing therapeutic hypothermia for hypoxic-ischemic encephalopathy will be enrolled in a new protocol that will allow mothers to hold their infants during the hypothermia treatment period. This is a safety study that will assess whether or not there is an increase in adverse event frequency in infants that are held during hypothermia. Parents and NICU nurses will be given a questionnaire after holding is complete investigating their feelings on maternal-infant bonding and safety of the holding protocol.

ELIGIBILITY:
Inclusion Criteria:

* Infant must have a gestational age of greater than or equal to 35 weeks
* Infant must be undergoing treatment with therapeutic hypothermia
* Infant must be without seizures in the first 24 hours of treatment based on EEG
* Infant must be clinically stable on bubble CPAP, nasal cannula, or no respiratory support.
* Informed consent must be signed by the mother at Maine Medical Center

Exclusion Criteria:

* Infant is intubated
* Infant is being treated with inhaled nitric oxide
* Presence of Persistent Pulmonary Hypertension of the Newborn
* Presence of seizure on EEG
* Use of vasopressors or paralytic agents
* Presence of chest tubes, wound vacuums, or drains
* Neonatal abstinence syndrome

Ages: 24 Hours to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-09-23 (Actual); Study Completion 2017-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexa Craig, MD, MSc, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Craig A, Deerwester K, Fox L, Jacobs J, Evans S. Maternal holding during therapeutic hypothermia for infants with neonatal encephalopathy is feasible. Acta Paediatr. 2019 Sep;108(9):1597-1602. doi: 10.1111/apa.14743. Epub 2019 Mar 5. PMID 30721531

RESULTS

PARTICIPANT FLOW:
Groups:
- Holding Group: Intervention was mothers being able to hold their infants for 30 minutes during therapeutic hypothermia. Inclusion criteria were gestational age at birth of 35 weeks or greater, absence of clinical or electrographic seizures during the first 24 hours of TH, and designation as "clinically stable" by the attending neonatologist with the infant on room air, nasal cannula, or continuous positive airway pressure (CPAP). Exclusion criteria were intubation, use of inhaled nitric oxide for persistent pulmonary hypertension of the newborn, presence of seizures on EEG, use of vasopressors or paralytic agents, presence of chest tubes, wound vacuums, or drains, and in utero opiate exposure. Written informed consent was obtained from the mother for all patients.
Period: Overall Study
Arm/Group | Holding Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Holding Group: Inclusion criteria were gestational age at birth of 35 weeks or greater, absence of clinical or electrographic seizures during the first 24 hours of TH, and designation as "clinically stable" by the attending neonatologist with the infant on room air, nasal cannula, or continuous positive airway pressure (CPAP). Exclusion criteria were intubation, use of inhaled nitric oxide for persistent pulmonary hypertension of the newborn, presence of seizures on EEG, use of vasopressors or paralytic agents, presence of chest tubes, wound vacuums, or drains, and in utero opiate exposure. Written informed consent was obtained from the mother for all patients.
Arm/Group | Holding Group
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events (Safety)
Description: Assess the frequency of adverse events during the holding intervention including unintentional rewarming of the infant, dislodged infant catheters (umbilical arterial/venous lines, urinary catheter, iv) or infant intolerance of holding due to vital sign instability.
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Holding Group
Number analyzed (Participants) | 10
Participants | 0

2. Secondary Outcome: Qualitative Experience of Mothers: Before I Could Hold my Baby, I Would Describe Our Ability to Bond as:
Description: A novel tool was developed to assess the mothers' subjective level of stress and bonding with her infant after holding by a questionnaire.
  1. Before I could hold my baby, I would describe our ability to bond as:
  1. Very easy to bond
  2. Easy to bond
  3. Hard to bond
  4. Very hard to bond
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Groups:
- Holding Group: Holding during cooling: An initial set of vital signs will be recorded before the infant is removed from the isolette. The mother will sit in a reclining chair next to the isolette and place a thermal barrier over her chest and abdomen. The infant will be transferred to the mother by placing the hands under the cooling blanket so as to move the infant and cooling blanket together as one unit. The mother will be allowed to hold
Arm/Group | Holding Group
Number analyzed (Participants) | 10
Participants
  Very easy to bond | 0
  Easy to bond | 2
  Hard to bond | 5
  Very hard to bond | 3

3. Secondary Outcome: Qualitative Experience of Mothers: After Holding my Baby, I Feel Our Bond is:
Description: A novel tool was developed to assess the mothers' subjective level of stress and bonding with her infant after holding by a questionnaire.
  2. After holding my baby, I feel our bond is:
  1. Much stronger
  2. Stronger
  3. No change
  4. Weaker
  5. Much weaker
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Holding Group
Number analyzed (Participants) | 10
Participants
  Much stronger | 6
  Stronger | 4
  No change | 0
  Weaker | 0
  Much weaker | 0

4. Secondary Outcome: Qualitative Experience of Mothers: Before Holding my Baby, my Stress Level Was:
Description: A novel tool was developed to assess the mothers' subjective level of stress and bonding with her infant after holding by a questionnaire.
  3. Before holding my baby, my stress level was:
  1. Very high
  2. High
  3. Low
  4. Very low
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Holding Group
Number analyzed (Participants) | 10
Participants
  Very high | 6
  High | 3
  Low | 1
  Very low | 0

5. Secondary Outcome: Qualitative Experience of Mothers: After Holding my Baby, I Feel:
Description: 4. After holding my baby, I feel:
  1. Much more stressed
  2. More stressed
  3. No change
  4. Less stressed
  5. Much less stressed
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Holding Group
Number analyzed (Participants) | 10
Participants
  Much more stressed | 0
  More stressed | 0
  No change | 0
  Less stressed Less stressed | 3
  Much less stressed | 7

6. Secondary Outcome: Qualitative Experience of Mothers: I am Glad I Had the Opportunity to Hold my Baby During Treatment With Hypothermia
Description: 5. I am glad I had the opportunity to hold my baby during treatment with hypothermia
  1. Strongly agree
  2. Agree
  3. Disagree
  4. Strongly disagree
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Holding Group
Number analyzed (Participants) | 10
Participants
  Strongly agree | 10
  Agree | 0
  Disagree | 0
  Strongly disagree | 0

7. Secondary Outcome: Qualitative Experience of Mothers: I Think Other Parents Would Benefit From Holding Their Babies During Treatment With Hypothermia, Provided They Are Medically Stable
Description: 6. I think other parents would benefit from holding their babies during treatment with hypothermia, provided they are medically stable
  1. Strongly agree
  2. Agree
  3. Disagree
  4. Strongly Disagree
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Holding Group
Number analyzed (Participants) | 10
Participants
  Strongly agree | 10
  Agree | 0
  Disagree | 0
  Strongly disagree | 0

8. Secondary Outcome: Qualitative Experience of Nurses: Therapeutic Hypothermia is Emotionally Challenging to the Parents of the Infant.
Description: A novel tool was developed by the investigator to assess the nurses' subjective level of comfort with mothers holding their infants during the cooling protocol.
  Therapeutic hypothermia is emotionally challenging to the parents of the infant.
  A. Strongly agree B. Agree C. Disagree D. Strongly Disagree
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Groups:
- Nursing Participation: Nurses responded to 16 question survey upon completion of holding.
Arm/Group | Nursing Participation
Number analyzed (Participants) | 8
Participants
  Strongly agree | 1
  Agree | 7
  Disagree | 0
  Strongly disagree | 0

9. Secondary Outcome: Qualitative Experience of Nurses: Treatment With Therapeutic Hypothermia Makes it Difficult for Parents to Bond With Their Infant.
Description: A novel tool was developed by the investigator to assess the nurses' subjective level of comfort with mothers holding their infants during the cooling protocol.
  Treatment with therapeutic hypothermia makes it difficult for parents to bond with their infant.
  A. Strongly agree B. Agree C. Disagree D. Strongly Disagree
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Participation
Number analyzed (Participants) | 8
Participants
  Strongly agree | 3
  Agree | 5
  Disagree | 0
  Strongly disagree | 0

10. Secondary Outcome: Qualitative Experience of Nurses: After Assisting With the Holding Protocol, the Mother's Emotional Response to Her Infant's Treatment is...
Description: A novel tool was developed by the investigator to assess the nurses' subjective level of comfort with mothers holding their infants during the cooling protocol.
  After assisting with the holding protocol, the mother's emotional response to her infant's treatment is...
  A. Strongly more positive B. More positive C. No change D. More negative E. Strongly more negative
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Participation
Number analyzed (Participants) | 8
Participants
  Strongly more positive | 5
  More positive | 1
  No change | 2
  More negative | 0
  Strongly more negative | 0

11. Secondary Outcome: Qualitative Experience of Nurses: After Seeing the Mother Hold Her Infant, the Maternal-infant Bond is a...
Description: A novel tool was developed by the investigator to assess the nurses' subjective level of comfort with mothers holding their infants during the cooling protocol.
  After seeing the mother hold her infant, the maternal-infant bond is a... A. Much stronger bond B. Stronger bond C. No change D. Weaker bond E. Much weaker bond
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Participation
Number analyzed (Participants) | 8
Participants
  Much stronger bond | 4
  Stronger bond | 2
  No change | 0
  Weaker bond | 2
  Much weaker bond | 0

12. Secondary Outcome: Qualitative Experience of Nurses: After Assisting With the Holding Protocol, I Feel That Holding During Cooling is Safe.
Description: A novel tool was developed by the investigator to assess the nurses' subjective level of comfort with mothers holding their infants during the cooling protocol.
  After assisting with the holding protocol, I feel that holding during cooling is safe.
  A. Strongly agree B. Agree C. Disagree D. Strongly disagree
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Participation
Number analyzed (Participants) | 8
Participants
  Strongly agree | 6
  Agree | 2
  Disagree | 0
  Strongly disagree | 0

13. Secondary Outcome: Qualitative Experience of Nurses: I Would Like to See Holding During Cooling Become a Standard Practice in Our NICU, so Long as the Infant is Otherwise Medically Stable.
Description: A novel tool was developed by the investigator to assess the nurses' subjective level of comfort with mothers holding their infants during the cooling protocol.
  I would like to see holding during cooling become a standard practice in our NICU, so long as the infant is otherwise medically stable.
  A. Strongly agree B. Agree C. Disagree D. Strongly disagree
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Participation
Number analyzed (Participants) | 8
Participants
  Strongly agree | 6
  Agree | 2
  Disagree | 0
  Strongly disagree | 0

14. Secondary Outcome: Qualitative Experience of Nurses: After Having Been Held, the Infant Has Become…
Description: A novel tool was developed by the investigator to assess the nurses' subjective level of comfort with mothers holding their infants during the cooling protocol.
  I would like to see holding during cooling become a standard practice in our NICU, so long as the infant is otherwise medically stable.
  A. Much easier to care for B. Easier to care for C. No change D. Harder to care for E. Much harder to care for
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nursing Participation
Number analyzed (Participants) | 8
Participants
  Much easier to care for | 1
  Easier to care for | 3
  No change | 4
  Harder to care for | 0
  Much harder to care for | 0

ADVERSE EVENTS:
Time Frame: Adverse events were tracked for the three days of therapeutic hypothermia.
Arm/Group | Holding Group
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT03079284/Prot_SAP_000.pdf